CLINICAL TRIAL: NCT03675997
Title: GRAFted Patients' anxieTY Report (GRAFTY)
Brief Title: GRAFted Patients' anxieTY Report
Acronym: GRAFTY
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0202; 2018-A02005-50 (Other: ANSM)
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Autologous Transplant Indication
Keywords: Autograft; Anxiety; Protected environment
MeSH Terms: conditions — Anxiety Disorders | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autografted patients: Patients hospitalized in the hematological department of the Institute will complete the first day of conditioning and then weekly HAD (Hospital Anxiety and Depression) scale.
  Interventions: Other: HAD (Hospital Anxiety and Depression) scale

INTERVENTIONS:
Other: HAD (Hospital Anxiety and Depression) scale — HAD (Hospital Anxiety and Depression) scale will be completed and reported by patients the first day of conditioning and then weekly from day 0 corresponding to the autograft, until their last day in the hematological department.

SUMMARY:
Autograft is a technique requiring several weeks of hospitalization in a protected environment and can be a source of anxiety of different natures for patients. In this study, level of anxiety will be reported weekly throughout hospitalizations for autologous transplant, to detect the most stressful period.

DETAILED DESCRIPTION:
Autograft is one of hematological malignancies treatment, such as lymphoma and myeloma. This technique requires several weeks of hospitalization in a protected environment and can be a source of anxiety of different natures for patients. According to the medical and scientific report of the Biomedicine Agency in 2016, 3 043 patients were involved in an autologous transplant, which represents a significant number of patients potentially exposed to these types of anxiety.

That is why it will be interesting in this study to report weekly the level of anxiety throughout their hospitalization for the autologous transplant, to detect the most stressful period.

A validated questionnaire will be used: the HAD (Hospital Anxiety and Depression) scale of anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Autograft indication according to the Multidisciplinary Concertation Meeting

Exclusion Criteria:

* Incapacity to complete surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for autograft will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
Anxiety and depression measure | 30 days
  The aim of this study is to measure patients anxiety and depression, using the HAD : Hospital Anxiety and Depression scale.
  Scores of the HAD scale can be defined as:
  * By adding the points of the answers: 1, 3, 5, 7, 9, 11, 13: we obtain the "Total A" which corresponds to the measure of the anxiety, then:
  * 7 or less: absence of symptomatology;
  * 8 to 10: doubtful symptomatology;
  * 11 and above: certain symptomatology.
  * By adding the points of the answers: 2, 4, 6, 8, 10, 12, 14: we obtain the "Total B" which corresponds to the measure of the depression, then:
  * 7 or less: absence of symptomatology;
  * 8 to 10: doubtful symptomatology;
  * 11 and above: certain symptomatology.
  The minimal score is 0 and the maximal total score is 42.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Morisson, MD, Principal Investigator — Institut de Cancérologie Lucien Neuwirth
Locations (1):
- Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez, France

IPD SHARING:
Plan to Share IPD: No